CLINICAL TRIAL: NCT00951626
Title: A Standardized Nursing Intervention Protocol for HCT Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 05081; R01CA107446 (NIH); P30CA033572 (NIH); CHNMC-05081; CDR0000643265 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2009-08-01; First posted 2009-08-04 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms; Psychosocial Effects of Cancer and Its Treatment; Therapy-related Toxicity
Keywords: psychosocial effects of cancer and its treatment; therapy-related toxicity; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult Hodgkin lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; recurrent mycosis fungoides/Sezary syndrome; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); atypical chronic myeloid leukemia, BCR-ABL negative; blastic phase chronic myelogenous leukemia; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; chronic eosinophilic leukemia; primary myelofibrosis; chronic neutrophilic leukemia; de novo myelodysplastic syndromes; myelodysplastic/myeloproliferative neoplasm, unclassifiable; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; refractory multiple myeloma
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Leukemia, Myeloid, Acute; Leukemia, Hairy Cell; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Neutrophilic, Chronic | interventions — Diet Therapy; Early Intervention, Educational; Peripheral Blood Stem Cell Transplantation; Psychiatric Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: exercise intervention — Those on the Standard Nursing Intervention Program will be offered six educational sessions spaced over the first 3 months after discharge.
  Those on the Usual Care plus Attention Control program will be offered a copy of the complete teaching manual for Hematopoietic Cell Transplant patients which will stay with them during hospitalization and be sent home after discharge.
Behavioral: telephone-based intervention — Those on the Standard Nursing Intervention Program will receive phone calls from the Intervention Nurse after the first 3 months and then monthly calls up to 12 months post hospital discharge.
  For those on the Usual Care plus Attention Control program, the Intervention Nurse will be available by phone or email within 48 hours of request for 100 days post transplant.
Dietary Supplement: dietary intervention — Those on the Standard Nursing Intervention Program will be offered six educational sessions spaced over the first 3 months after discharge.
  Those on the Usual Care plus Attention Control program will be offered a copy of the complete teaching manual for Hematopoietic Cell Transplant patients which will stay with them during hospitalization and be sent home after discharge.
Other: educational intervention — Those on the Standard Nursing Intervention Program will be offered six educational sessions spaced over the first 3 months after discharge.
  Those on the Usual Care plus Attention Control program will be offered a copy of the complete teaching manual for Hematopoietic Cell Transplant patients which will stay with them during hospitalization and be sent home after discharge.
Other: questionnaire administration — For both groups of participants, administered at baseline (prior to hospital discharge and 3, 6, and 12 months post hospital discharge.
Procedure: allogeneic bone marrow transplantation — Patient with a diagnosis of a hematologic cancer scheduled for a single allogeneic bone marrow transplant.
Procedure: allogeneic hematopoietic stem cell transplantation — Patient with a diagnosis of a hematologic cancer scheduled for a single allogeneic stem cell transplant.
Procedure: assessment of therapy complications — Collected throughout the 12 month study period
Procedure: peripheral blood stem cell transplantation — Patient with a diagnosis of a hematologic cancer scheduled for a single allogeneic stem cell transplant.
Procedure: psychosocial assessment and care — Those on the Standard Nursing Intervention Program will be offered six educational sessions spaced over the first 3 months after discharge. They will also receive phone calls from the Intervention Nurse after the first 3 months and then monthly calls up to 12 months post hospital discharge.
Procedure: quality-of-life assessment — For both groups of participants, questionnaires administered at baseline (prior to hospital discharge and 3, 6, and 12 months post hospital discharge.
Procedure: standard follow-up care — Those on the Usual Care plus Attention Control program will be offered a copy of the complete teaching manual for Hematopoietic Cell Transplant patients which will stay with them during hospitalization and be sent home after discharge. Also the Intervention Nurse will be available by phone or email within 48 hours of request for 100 days post transplant.

SUMMARY:
RATIONALE: Visiting patients at home to teach them about self care after a stem cell transplant may be more effective than standard therapy in improving quality of life.

PURPOSE: This clinical trial is studying home visits to see how well they work compared with standard therapy in treating patients undergoing donor stem cell transplant for hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Test the effects of a Standardized Nursing Intervention Protocol (SNIP) on overall quality of life (QOL); physical, psychological, social, and spiritual well-being subscales; and functional status of patients undergoing allogeneic hematopoietic stem cell transplantation (AHSCT) at discharge, 3, 6, and 12 months post-hospitalization as compared to AHSCT patients who receive the usual care and attention control.

Secondary

* Test the effects of SNIP-AHSCT on time-to-first complication, total number of complications, and mortality across these groups of patients.
* Identify subgroups of patients who benefit most from the SNIP-AHSCT in relation to sociodemographic characteristics, disease and clinical factors, and transplant factors.
* Decompose the effect of the SNIP-AHSCT on QOL into direct and indirect effects.

OUTLINE: Patients are randomized to 1 of 2 treatment groups.

* Group 1: Patients receive home teaching visits on medical aspects of self care, monitor and respond to signs and symptoms of infections, recommended exercise and nutrition program, relevant literature on bone marrow transplantation, diet, nutrition, and a variety of resources at 1, 2, and 3 months after hospital discharge. Patients also receive telephone-reinforcement calls monthly in months 4-12, and have a 24-hour telephone availability throughout the study. Patients complete the City of Hope quality of life questionnaires on physical, psychological, social, and spiritual well-being, and physical functional status at discharge, and then at 3, 6, and 12 months after hospitalization.
* Group 2: Patients receive usual medical care and attention at discharge, and then at 3, 6, and 12 months after hospitalization. Patients also have a hot-line availability throughout the study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of a hematologic cancer (e.g., leukemia or lymphoma)
* Scheduled for a single allogeneic bone marrow or peripheral blood stem cell transplantation

PATIENT CHARACTERISTICS:

* Living within a 50-mile radius of the City of Hope National Medical Center
* English-speaking

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior hematopoietic stem cell transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2005-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Overall quality of life (physical, psychological, social, and spiritual well-being) | Baseline (discharge from hospital following Hematopoietic Cell Transplant) and 3, 6, and 12 months post baseline
Functional status | Baseline (discharge from hospital following Hematopoietic Cell Transplant) and 3, 6, and 12 months post baseline

SECONDARY OUTCOMES:
Time-to-first complication | Baseline (discharge from hospital following Hematopoietic Cell Transplant) and 3, 6, and 12 months post baseline
Total number of complications | Baseline (discharge from hospital following Hematopoietic Cell Transplant) and 3, 6, and 12 months post baseline
Mortality | Baseline (discharge from hospital following Hematopoietic Cell Transplant) and 3, 6, and 12 months post baseline

CONTACTS AND LOCATIONS:
Overall Officials: Marcia Grant, RN, DNSc, FAAN, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States